CLINICAL TRIAL: NCT06185621
Title: The Effect of 100mg Aspirin on Recurrent Acute Pancreatitis: a Prospective Cohort Study
Brief Title: The Effect of Aspirin on Recurrent Acute Pancreatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KY20232303-F-1
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Acute Pancreatitis; Prevention; Aspirin
MeSH Terms: conditions — Pancreatitis | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Patients received oral 100mg aspirin, one tablet daily for 2 years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 100mg aspirin group (Experimental): Patients received oral 100mg aspirin, one tablet daily for 2 years
  Interventions: Drug: 100mg aspirin

INTERVENTIONS:
Drug: 100mg aspirin — Patients received oral 100mg aspirin, one tablet daily for 2 years

SUMMARY:
Recurrent acute pancreatitis (RAP) was defined as two or more occurrences of acute pancreatitis, which was associated with higher percentages of morbidities and mortalities, lower patients' life quality and increased health-care costs. Current interventions, including cholecystectomy and abstain from drinking were reported to be effective methods for preventing the recurrences of biliary and alcoholic etiologies, respectively. However, there were no effective preventions for other etiologies, such as idiopathic etiologies. Non-steroid anti-inflammatory drugs (NSAIDs), including indomethacin, diclofenac and aspirin could inhibiting the inflammatory cascade of pancreatitis. In this study, we aimed at exploring the effects of 100mg aspirin on reducing the occurrences of recurrent acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with with recurrent acute pancreatitis

Exclusion Criteria:

* Less than 2 episodes of acute pancreatitis in the past year
* Latrogenic AP (pancreatitis due to endoscopic retrograde cholangiopancreatography, surgery, or after other invasive treatment). Iatrogenic pancreatitis will not count as an episode of recurrent pancreatitis
* Previous allergy to Non-Steroid Anti-inflammatory Drugs (NSAIDs)
* Regularly taking aspirin or other NSAIDs >3 doses per week
* Contradictions for the medications of NSAIDs, including Active peptic ulcer disease or gastrointestinal hemorrhage within 3 months or previous peptic ulcer, history of significant hepatic or renal disease, platelet count less than 100X10^9/L or international normalized ratio (INR) >1.5)
* Biliary stones
* Receiving endoscopic sphincterotomy and/or pancreatic stent placement and/or cholecystectomy and/or pancreatic surgery after the latest pancreatitis or planning to undergo one of those interventions within preceding 2 years
* Patients with the level of serum triglycerides of >5.65 mmol/L and did not receive regular lipid-lowering therapy
* Primary hyperparathyroidism has been well-treated after last episode of pancreatitis and recruitment or will be operated in <2 years
* Patients with previously heavy alcohol consumption (50g/day for men, 40g/day for women) and have not quit drinking, or have significant withdrawal symptoms
* Pregnant or breastfeeding patients
* Inability to give informed consents

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
The mean interval between two consecutive occurrences of acute pancreatitis during follow-up | 2 years
  Acute pancreatitis was defined as meeting two or three following items: (1) acute onset of a persistent, severe, epigastric pain often radiating to the back. (2) Serum amylase and/or lipase concentrations at least three times higher than upper limit of normal value. (3) Abdominal imaging examination results showed pancreatic inflammation.

SECONDARY OUTCOMES:
The numbers of acute pancreatitis during follow-up | 2 years
The numbers of pancreatitis with different severity evaluated by revised Atlanta criteria | 2 years
  Mild acute pancreatitis, no organ failure and no local or systemic complications; Moderately severe acute pancreatitis, organ failure that resolves within 48 h (transient organ failure) and/or Local or systemic complications without persistent organ failure.
  Severe acute pancreatitis, Persistent organ failure (>48 h).
The hospitalization days due to acute pancreatitis | 2 years
The rate of patients with chronic pancreatitis. | 2 years
  chronic pancreatitis was defined according to the Asia&Pacific consensus report, when meeting one of the following conditions: (1) pancreatic calcification on cross-sectional imaging; (2) pancreatic ductal changes on endoscopic retrograde cholangiopancreatography (ERCP); (3) abnormal pancreatic function test results; (d) confirmed CP on endoscopic ultrasound; and (4) histological evidence of CP.
The rate of patients with new-onset diabetes | 2 years
The numbers of aspirin tablets the patients actually take | 2 years
The mortality rate | 2 years
The rate of patients who had adverse events due to oral aspirin | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Air Force Military Medical University, China, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Sankaran SJ, Xiao AY, Wu LM, Windsor JA, Forsmark CE, Petrov MS. Frequency of progression from acute to chronic pancreatitis and risk factors: a meta-analysis. Gastroenterology. 2015 Nov;149(6):1490-1500.e1. doi: 10.1053/j.gastro.2015.07.066. Epub 2015 Aug 20. PMID 26299411
- [Background] Guda NM, Muddana V, Whitcomb DC, Levy P, Garg P, Cote G, Uc A, Varadarajulu S, Vege SS, Chari ST, Forsmark CE, Yadav D, Reddy DN, Tenner S, Johnson CD, Akisik F, Saluja AK, Lerch MM, Mallery JS, Freeman ML. Recurrent Acute Pancreatitis: International State-of-the-Science Conference With Recommendations. Pancreas. 2018 Jul;47(6):653-666. doi: 10.1097/MPA.0000000000001053. PMID 29894415
- [Background] Takada Y, Bhardwaj A, Potdar P, Aggarwal BB. Nonsteroidal anti-inflammatory agents differ in their ability to suppress NF-kappaB activation, inhibition of expression of cyclooxygenase-2 and cyclin D1, and abrogation of tumor cell proliferation. Oncogene. 2004 Dec 9;23(57):9247-58. doi: 10.1038/sj.onc.1208169. PMID 15489888